CLINICAL TRIAL: NCT06681350
Title: Evaluation of Diagnostic Effectiveness and Reliability of a Telemedical Examination with Occyo One Vs Traditional Slit Lamp-based Examination After Cataract Surgery
Brief Title: Occyo Tele-ophthalmology Study
Acronym: OTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OTS
Record Dates: First submitted 2024-09-12; First posted 2024-11-08 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cataract
Keywords: Cataract; Slit lamp; Telemedical examination; Image based diagnosis
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Occyo One Anterior Segment Imaging (Other): Imaging of the anterior segment of the eye for telemedical assessment.
  Interventions: Device: Ocular surface imaging

INTERVENTIONS:
Device: Ocular surface imaging — Telemedical examination of high-resolution, all-in-focus images of the cornea, sclera, conjunctiva, and lid margins for montioring of postoperative complications

SUMMARY:
The prospective, (observer) blinded clinical trial at the University Hospital for Ophthalmology includes patients routinely scheduled for cataract surgery at the Medical University of Innsbruck.

Patients are enrolled one week prior to their planned cataract surgery. The participants will undergo a screening in which, in addition to the ophthalmological standard examinations, Occyo One images of the anterior segment of the eye are taken. After surgery, a post-operative follow-up visit takes place and a second set of Occyo One images will be generated.

During the postoperative check-up, the study team at the trial center decides-based on defined criteria (medical history, slit lamp examination results)-whether a change in the subsequent patient management is necessary due to the presence of postoperative complications (unexpected management changes = UMC).

Up on completion of all patient visits/study-specific measurements and data collection, information regarding diagnostic criteria and the Occyo One images are sent to an external, blinded ophthalmologist for telemedical assessment. Based on the available information and images, the blinded ophthalmologist decides whether a change in patient management should have been made or not.

The difference in the detection of an event resulting in a UMC is the primary objective of this clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Understands and agrees to comply with the study procedures and provides written informed consent as documented by signature
2. Patients scheduled to undergo cataract surgery
3. Male or female patient aged ≥ 50 years at time of consent

Exclusion Criteria:

1. Woman of childbearing potential (WOCBP)

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Unexpected Management Changes | 1 week
  Difference of the detection rate of postoperative complications of cataract surgery defined as any event requiring unexpected management changes (UMC) comparing physical slit lamp examination to independent Occyo One image-based telemedical diagnosis by a blinded examiner.

SECONDARY OUTCOMES:
Efron Grading | 1 week
  Difference among Efron Grading for ocular redness, derived from physical slit lamp examination versus blinded image-based telemedical assessment of Occyo One photographs. Correlation of Efron Grading of conjunctival redness with objective anterior chamber laser flare photometry.
Oxford Cataract Treatment and Evaluation Team (OCTET) Grading of corneal edema | 1 week
  Difference among OCTET grading of corneal edema derived from physical slit lamp examination versus blinded image-based telemedical assessment of Occyo One photographs.
  Grade Severity Description
  1. mild Transient corneal edema
  2. moderate Transient corneal edema with Descemet's membrane folds of <10
  3. severe Transient corneal edema with Descemet's membrane folds of >10
National Eye Institute (NEI) Grading Scale | 1 week
  Difference among NEI grading score for corneal fluorescein staining derived from physical slit lamp examination versus blinded image-based telemedical assessment of Occyo One photographs.
  Each of the 5 areas of the corneal surface are scored and summed to a total score (Grade 0-3).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, University Hospital for Ophthalmology and Optometry, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No